CLINICAL TRIAL: NCT02286011
Title: Phase I Clinical Trial on Intramuscular Infusion of Autologous Bone Marrow Stem Cells in Patients With Amyotrophic Lateral Sclerosis.
Brief Title: Intramuscular Infusion of Autologous Bone Marrow Stem Cells in Patients With Amyotrophic Lateral Sclerosis
Acronym: TCIM/ELA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Spanish National Health System (Other); Hospital Universitario Virgen de la Arrixaca (Other); Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other); Public Health Service, Murcia (Other); Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCIM/ELA; 2011-004801-25 (EudraCT Number)
Record Dates: First submitted 2014-10-24; First posted 2014-11-07 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MNC (Mononuclear cells) (Experimental): All patients included in the clinical trial will receive an intramuscular infusion of autologous mononuclear cells (MNC) of Bone Marrow (BM) in TA muscle of one of the lower limb (experimental group). The lower limb on the CMN infuse autologous BM will be determined randomly.
  The average dose is 550 millions of cells (100-1200 million) diluted in 2 ml. saline
  Interventions: Biological: MNC (Mononuclear cells)
- Saline (Placebo Comparator): All patients included in the clinical trial will receive an intramuscular infusion of 2 mL of saline (placebo) in the TA muscle of the contralateral limb (group control).
  Interventions: Other: Saline

INTERVENTIONS:
Biological: MNC (Mononuclear cells) — The cells are infused into the TA muscle of the lower limb randomized as Group A (experimental) intramuscularly. The infusion is made with a needle, 26 gauge, at 4 points of the TA muscle a specific depth given by the neurophysiological study. The total volume infused will be 2 ml, 0.5 ml at each point.
  For infusion is as painless as possible for the patient to comply exactly with stereotactic indications of neurophysiology, the infusion was made at a uniform controlled rate and for this, the syringe is placed on a Yesargil arm, equipped with a microinjector and controlled infusion device.
  Arms: MNC (Mononuclear cells)
Other: Saline — The placebo, 2ml of saline, will be infused like in the experimental arm.
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety of Intramuscular Infusion of Autologous Bone Marrow Stem Cells in Patients With Amyotrophic Lateral Sclerosis by a prospective, single-center, randomized, parallel, double-blind, placebo-controlled phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or probable ALS according to the criteria established by the World Federation of Neurology
* Patient that provides reasonable assurance of adherence to protocol.
* Neurophysiological data confirming affectation of lower motor neurons in the lumbar region.
* Assessment of motor deficits in dorsiflexion of both feet (4 or 5 points on the MRC scale)
* The patient must fulfill all inclusion criteria.

Exclusion Criteria:

* Diabetes Mellitus.
* Other diseases that may present with polyneuropathy.
* Previous history of stroke.
* Prior Pathology of the peripheral nervous system affecting one or both lower limbs with or without clinically evident neurological sequelae.
* Pregnant or breastfeeding patients active.
* Patients physiologically capable of becoming pregnant, unless they are using reliable contraception.
* Patients with cardiac disease, renal, hepatic, systemic, immune that may influence patient survival during the test.
* Positive serology for hepatitis B, hepatitis C or HIV.
* Clinical and anesthesiologic Criteria, contraindicating either sedation or extraction of MO (Altered coagulation system or anticoagulated patient with inability to withdraw anticoagulation, hemodynamic instability, altered skin puncture site, etc.)
* Included in other clinical trials in the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of serious and non-serious adverse events related to the use of bone marrow mononuclear cells in patients with Amyotrophic Lateral Sclerosis. | 24 months from baseline

SECONDARY OUTCOMES:
Estimated number of motor units (MUNE) | 24 months from baseline
  Several techniques for estimating the MUNE, all based on the relationship between the amplitude or area of compound muscle action potential (CMAP) and amplitude or area corresponding to a single motor unit response. The differences between the techniques are due to the different ways of estimating the amplitude of the responses for individual motor units. The study will use two techniques:
  Incremental Technique: The unitary amplitude (or area) of individual motor units are calculated from the responses to increasing intensities stimuli near of intensity threshold (Dantes and McComas, 1991) Statistical technique: The unit amplitude (or area) of the individual motor units are calculated from the amplitude variations (or area) of the muscle action potential obtained in response to stimuli from a fixed intensity (Daube, 2006)
Compound muscle action potential (CMAP) | 24 months from baseline
  CMAP is registered after supramaximal stimulation intensity (0.1-0.2 ms pulses at 1 Hz) of the common peroneal nerve at the level of the head of the fibula. The electrical stimulus is placed in a fixed position during the entire registration process. CMAP will be recorded simultaneously in 5 positions along longitudinally oriented TA muscle. To determine these 5 positions bony landmarks that are reproducible between members and between different patients will be used.
Fiber density (FD) | 24 months from baseline
  Quantifies the average number of muscle fibers per motor unit. It is obtained from single fiber recordings made with electrodes. The average number of motor unit potentials is calculated in 20 different positions in the muscle.
Muscle force MRC (Medical Research Council) score | 24 months from baseline
Maximum force developed in an isometric contraction of the tibialis anterior (TA) muscle. | 24 months from baseline
  The measurement will be done in Newtons, with a dynamometer during dorsiflexion of the foot (from certain angles).
Maximum transversal area of the tibialis anterior (TA) | 24 months from baseline
  The area will be measured in cm2 by echography.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín A Gómez Espuch, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Clinical Universitary Hospital Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- [Result] Blanquer M, Moraleda JM, Iniesta F, Gomez-Espuch J, Meca-Lallana J, Villaverde R, Perez-Espejo MA, Ruiz-Lopez FJ, Garcia Santos JM, Bleda P, Izura V, Saez M, De Mingo P, Vivancos L, Carles R, Jimenez J, Hernandez J, Guardiola J, Del Rio ST, Antunez C, De la Rosa P, Majado MJ, Sanchez-Salinas A, Lopez J, Martinez-Lage JF, Martinez S. Neurotrophic bone marrow cellular nests prevent spinal motoneuron degeneration in amyotrophic lateral sclerosis patients: a pilot safety study. Stem Cells. 2012 Jun;30(6):1277-85. doi: 10.1002/stem.1080. PMID 22415951
- [Derived] Geijo-Barrientos E, Pastore-Olmedo C, De Mingo P, Blanquer M, Gomez Espuch J, Iniesta F, Iniesta NG, Garcia-Hernandez A, Martin-Estefania C, Barrios L, Moraleda JM, Martinez S. Intramuscular Injection of Bone Marrow Stem Cells in Amyotrophic Lateral Sclerosis Patients: A Randomized Clinical Trial. Front Neurosci. 2020 Mar 24;14:195. doi: 10.3389/fnins.2020.00195. eCollection 2020. PMID 32265627